CLINICAL TRIAL: NCT06777693
Title: The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Older Adults: a Feasibility Study
Acronym: UPS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NKS Olaviken Gerontopsychiatric Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 769706
Record Dates: First submitted 2024-09-30; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Emotional Disorders
Keywords: Emotional disorders; Anxiety; Depression; Avoidant coping; Neuroticism
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study aims to investigate the feasibility of the Unified Protocol for old adults (older than 65) in an outpatient clinic in terms of the four aspects; acceptance and percieved helpfulness, practical feasibility, reliable change and iterative modifications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Other): The treatment follows the translation of the Danish manual of the group version of UP, with 12 group sessions. Each group will consist of up to eight participants, and two therapists trained in UP. Diagnostic assessment and screening are conducted in the clinic before inclusion, but one session is reserved for baseline assessment and neuropsychological testing before participating in the intervention. Initially, the participants will have two individual sessions, including the case formulation and the goal-setting session of UP. Then, the participants will undergo the Unified Protocol in a group format, consisting of weekly sessions over 11 weeks and a booster session after one month. Post-assessment is conducted within the first 14 days after the last group session.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol group format involves 12 sessions focusing on goal setting and motivation, understanding emotions, mindful emotion awareness, cognitive flexibility, countering emotionat behaviours, understanding and confronting physical sensations, emotion exposure and relapse prevention.
  The UP model directly approaches the patient's emotion regulation by focusing on cognitive flexibility, exposure exercises, mindful awareness, acceptance, and other evidence-based therapeutic approaches known from cognitive-behavioural therapy (CBT), emotion-focused therapy (EFT) and mindfulness-based interventions.

SUMMARY:
Psychological treatment is less likely to be offered in an older population. In order to adapt treatment effectively for this population, more research is necessary. This study will investigate the feasibility of Unified Protocol Senior (65 years and older) in a group format. Patients with emotional disorders (i.e. anxiety or depression) is offered diagnostic and cognitive evaluations, two individual sessions and twelve group sessions lasting 2 hours. The participants psychological symptoms will be examined pre-, during- and post-treatment. Qualitative interviews will be conducted after treatment in order to understand the participants experience of and outcome of the treatment. The study will investigate whether any unwanted experiences occurred during treatment.

The study is planning on carrying out four seperate treatmentgroups consisting of 6-8 patients. Information gathered from one group will be used to adapt the group sessions for the consecutive treatment group. This will be done until a feasible format is reached.

DETAILED DESCRIPTION:
Emotional disorders such as anxiety and depression are the most common mental health problems affecting older people, and are highly comorbid . The prevalence is high (greater than 25 %), with increasing prevalence for people with comorbid somatic disorders (greater than 40%). Evidence suggests that psychological treatment for older adults is as effective as for working-age adults and maybe even more effective in old adults with comorbid somatic disorders. Despite this, older adults are generally under-represented in psychological services.

Most older adults with emotional disorders receive psychopharmacological treatment as the first choice, even when national and clinical guidelines suggest offering psychological treatment as a first choice or combining medication and psychological treatment. Studies show that adults older than 65 prefer psychological therapy over psychotropic medication. Choosing psychological treatment also decreases risks associated with polypharmacy. Evidence shows that psychological treatment for common mental health problems in people older than 65 is effective. Implementing effective and available psychological treatment for people older than 65 in Norway is challenging, primarily due to lack of referral to mental health care units despite the guidance of priority for public mental health services recommend stressing the severity of symptoms and not age itself. Negative consequences for untreated mental health problems in older adults can have significant consequences on overall well-being, ranging from social isolation, cognitive decline, increased risk of suicide and exacerbating existing medical conditions. Thus, making evidence-based psychological services available for older adults is a highly relevant goal to achieve.

A key barrier challenging the implementation of evidence-based psychological treatment is that implementing diagnosis-specific protocols is not very well suited to the clinical settings where comorbidity and complexity are the norm. This is not specific for mental health care for people older than 65, implementing evidence-based psychological treatment is challenging in the health care systems in general. Accordingly, transdiagnostic treatment protocols have been developed over the last decades, where the treatment model targets underlying processes and mechanisms across different, but commonly comorbid, diagnoses. Barlow and colleagues have developed the "Unified protocol for transdiagnostic treatment of emotional disorders" in response to this issue. The Unified Protocol (UP) has shown promising results in treating anxiety and depression in various populations. However, its efficacy in older adults (older than 65 years) remains understudied. This is not specific to UP; most treatment protocols and outcome scales used in mental health care for adults are mainly developed for adults of working age and not adapted for the specific issues in late adulthood where immobility and social isolation, comorbid somatic disorders, and impaired executive functioning are more common. Given that psychological treatments for common mental health problems in people older than 65 are effective when adjusted to the needs of the population, investigating the feasibility of transdiagnostic treatments such as UP seems highly relevant. UP's theoretical foundations for development and maintenance of emotional disorders also seems transferable to our specific population, as described in the following section.

The transdiagnostic model of Unified Protocol According to UP, a typical shared personality dimension or temperament of people with emotional disorders is the vulnerability dimension of neuroticism, contributing to experience negative emotions with high intensity. People high in neuroticism tend to perceive these emotions as highly uncontrollable and dangerous, something that should be avoided. In sum, these negative emotions place the person at risk for persistent mental health problems. Two central processes may then contribute to the development of emotional disorders such as anxiety or depression. The first is the tendency to react aversively to intense emotional experiences. The second is the tendency for avoidant coping. UP targets both the vulnerability dimension of neuroticism and the dysfunctional coping of strong emotions. Further, the UP model directly approaches the patient's emotion regulation by focusing on cognitive flexibility, exposure exercises, mindful awareness, acceptance, and other evidence-based therapeutic approaches known from cognitive-behavioral therapy (CBT), emotion-focused therapy, and mindfulness-based interventions. Patients learn to understand their emotional experiences, observe them without judgment, stop avoidant coping, and change their behaviour toward reaching their goals. Avoiding negative stimuli is a common coping strategy for emotion regulation in old adults, but not all stressors may be avoided. Thus, learning to cope with emotional experiences through exposure as the theoretical foundation of UP suggests, seems transferable to our population. Clinical guidelines on emotional disorders, anxiety and depression in old adults also stress increasing the level of activity and break social isolation as important goals of treatment. Even if neural deterioration will occur with age, there is a potential of neuroplasticity and participants may still learn new behaviours and change in response to new experiences. However, identifying the older patient that will benefit from UP will probably require a wider initial assessment of cognitive functions (memory and executive function) and somatic condition (pharmacological treatment and somatic disorders potentially presenting as psychiatric symptoms).

Objectives UP has been investigated in large trials with promising results. A 14- session Group-based UP is currently implemented, and its feasibility is systematically evaluated in Norway in an adult population (18-40 years). There is an increasing expertise in western Norway on the method. There are also clinical experiences with an eight-session group based UP with older adults from a Geriatric Psychiatric Clinic (Äldrepsykiatrisk mottagning), Sahlgrenska Universitetssjukhuset (Gothenburg, Sweeden) where one found some effect on depressive symptoms and anxiety. Foremost, the participants with the best treatment effect changed the way they related to their thoughts and feelings (their psychological flexibility). As one participant said:" I can recognize my weak spots better. That is a window for change. When I recognize the patterns that are bad for me, it gives me the possibility to change them. I have learned a lot about emotions. I understand so much more, I recognize things that are not helpful to me." Experiences from these groups led the therapists to adapt the original manual and use less worksheets, practice mindful emotion awareness throughout the treatment, adjust psychoeducation to older adults' experiences, and adjust examples in the worksheets to older adults (less work, school and family-oriented examples).

Hence, the timing for testing UP in old adults in a research project seems optimal, with the possibility of collaborating with experienced clinicians and researchers in our project. This research proposal may well provide valuable insights into the feasibility of the Unified Protocol for treating emotional disorders in older adults. The findings will contribute to the growing body of evidence on transdiagnostic treatments and inform the development of adapted interventions for this population. The results will also inform the possibility of conducting a larger RCT with tailored treatment with UP for old adults on a later stage.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant symptoms of anxiety or depression based on self-report and clinical interview
* Score on the MMSE-NR above 26 and competent to give informed consent as evaluated by a structural clinical assessment
* Stable use of psychotropic medication for the last month. Periodic use of z-hypnotics is not exclusion criteria but will be restricted to a limited and pre-planned dosage per week. Stabilization of psychotropic medication can be offered to eligible patients before participation.
* Prepared to share their challenges and work on maladaptive emotion regulation strategies in a group setting.
* Able to attend most sessions.

Exclusion Criteria:

* Conditions requiring specialized treatment such as active psychosis and/or mania, untreated or unstable bipolar disorder, psychosis spectrum disorders or severe depressive episode
* Acutely increased risk of suicide or deliberate self-harm
* Dementia or amnestic mild cognitive impairment
* Substance abuse including psychoactive drugs
* Habitual use of prescribed anxiolytics or opiods. Help with gradual reduction and elimination before inclusion in treatment will be offered to potential participants
* Uncorrected hearing loss
* Symptoms of personality disorders that hinder participation in the group
* Simultaneously participating in other psychotherapy
* Living with ongoing highly social burden where greater flexibility in treatment is needed

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews | Immediately after the intervention
  Qualitative interviews relating to implementation, service and client outcomes will be conducted after the group treatment has finished. The interviews will focus on the participants experience with the feasibility of the interventions, especially regarding acceptability and adaptation as defined by Bowen and colleagues (2009).
Overall well-being | Baseline, and immediately after the intervention
  We use the World Health Organization Well-Being Index-5 (WHO-5, Topp et al., 2015) to measure overall subjective well-being. Scores range from 0-25 where higher scores indicate more well-being.
Geriatric Anxiety Inventory (GAI) | Baseline, after six weeks and immediately after the intervention
  Questionaire used to measure anxiety symptom severity in older adults. Higher scores (from 0-20) indicate higher symptom severity.
Generalized Anxiety Disorder Questionaire (GAD-7) | Baseline, after six weeks and immediately after the intervention
  Questionaire used to measure symptoms of generalized anxiety. Scores range from 0-21 where higher scores indicate higher symptom severity. The questionaire also ask how much these symptoms impact the persons ability to fuction effectively in every day activities.
Montgomery And Åsberg Depression Rating Scale (MADRS) | Baseline, after six weeks and immediately after the intervention
  Questionaire used to examine symptoms of depression as well as the severity of the symptoms. Scores range from 0-60 where higher scores indicate more depressive symptoms
Credibility/Expectancy Questionaire (CEQ) | Baseline, after six weeks and immediately after the intervention
  Test the participants expectancy and believes on whether the treatment will be helpful. Scores range from 6-51 where higher scores indicate higher beliefs and expectancy that the treatment will be helpful.
Overall Depression Severity and Impairment Scale (ODSIS) | Weekly, before every session for 12 weeks
  Questionaire developed as part of the UP manual used to track depression symptoms and their effect on function. Scores range from 0-20 where higher scores indicate higher symptom severity.
Overall Anxiety Severity and Impairment Scale (OASIS) | Weekly, before every session for 12 weeks
  Questionaire developed as part of the UP manual used to track anxiety symptoms and their effect on function. Scores range from 0-20 where higher scores indicate higher symptom severity.
The Norwegian Acceptance and Action Questionnaire version 2 (NAAQ-2) | Baseline, after six weeks and immediately after the intervention
  Measure the psychological flexibility of the participants. Higher scores (range 7-49) indicate lower levels of cognitive flexibility.
Negative Effects Questionnaire (NEQ) | Immediately after the intervention
  After the treatment, the participants are assessed using the Negative Effects Questionnaire to detect any adverse effects of the psychotherapy. These will be triangulated with the results from qualitative interviews assessing the experiences of the treatment. The scores is not numerical, but detects and describes any potential negative events from the treatment.
GeneActive Actigraph | During week 1, week 6 and week 12 of treatment procedure
  To register the participants' sleep and the 24-hour rest-activity-rhythm, we will use actigraphy. The actigraph (GeneActive) has been validated for use in older adults. It will be placed on the participants' non-dominant wrist.
The National Adult Reading Test (NART) | At baseline and immediately after the intervention
  Measure of general intelligence shown to correlate highly with premorbid intelligence. Scores range from 0-50 and will be reported as predicting premorbide intelligence below the average, on the average or above the average.
20 questions | Baseline, and immediately after the intervention
  The ability of abstract thinking and cognitive flexibility is assessed using 20 questions from Delis Kapln Executive Function system. Scores are reported as scaled scores below average, on average or above average.
Stroop test | Baseline, and immediately after the intervention
  Assesses the participants skills of inhibition. The scores are reported as scaled scores below average, on average or above average.
Numbers from WAIS-IV | Baseline, and immediately after the intervention
  Numbers from the Wechsler Adult Intelligence Scale will be used to assess the participants working memory. Scores are reported as scaled scores below average, on average or above average.
Trail Making Test B (TMT-B) | Immediately after the intervention
  TMT-B is used in the post-treatment measure, assessing cognitive shifting and psychomotoric tempo. Scales are reported as t-scores which fall below average, on average or above average.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine G Madsø, Clinical Psychology (PhD), Principal Investigator — NKS Olaviken Gerontopsychiatric Hospital
Locations (1):
- NKS NKS Olaviken Gerontopsychiatric Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow DH, Allen LB, Choate ML. Toward a Unified Treatment for Emotional Disorders - Republished Article. Behav Ther. 2016 Nov;47(6):838-853. doi: 10.1016/j.beth.2016.11.005. Epub 2016 Nov 10. PMID 27993336
- [Background] Braun, V., Clarke, V., Hayfield, N., Terry, G. (2019). Thematic analysis. In Handbook of Research Methods in Health Social Sciences (pp. 843-860). Springer.
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699